CLINICAL TRIAL: NCT06685406
Title: The Validity of Thorathic Fluid Content as Non Invasive Predictor on Weaning of Mechanical Ventilation in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Other Study IDs: 642/8 sep-2024
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2024-09

CONDITIONS: Cardiometry; Thorathic Fluid Content; Weaning From Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ventilated patients group
  Interventions: Diagnostic Test: Thorathic fluid content measurement by cardiometry

INTERVENTIONS:
Diagnostic Test: Thorathic fluid content measurement by cardiometry — Thorathic fluid content measurement by using cardiometry

SUMMARY:
Introduction Weaning from mechanical ventilation (MV) could be described as the process of removing ventilator support. Weaning from MV often implies two separate but closely linked views of care, elimination of MV of any artificial airway. Weaning from mechanical ventilation is a challenging step during recovery from critical illness (1).

Earlier patient weaning from mechanical ventilation is recommended to avoid complications of prolonged mechanical ventilation; however, premature weaning might result in extubation failure which is associated with poor outcomes (2).

The first step in weaning process is screening patients for readiness to be weaned from mechanical ventilation followed by the spontaneous breathing trial (SBT) by checking various indices carefully before starting SBT to ensure adequate oxygenation, ventilation, and airway reflexes (3).

However, a percent of patients fail and are re-intubated despite fulfillment of all the current weaning criteria and this may be due to the heterogeneity of critically ill patients which impairs the predictive accuracy of the available indices in different patient subgroups (4).

Various measures had been previously reported for evaluation of volume status such as fluid balance and echocardiography before the SBT aiming to identify patients who would benefit from diuretic therapy to achieve successful weaning from mechanical ventilation (5).

Nowadays, there is an increasing interest in cardiac factors, such as lung congestion and hypervolemia, as contributing elements in weaning failure and that needs expert physician such as echocardiography (6). So thoracic fluid content measurement may also be beneficial, more accurate and could give us a good idea about weaning of patients from mechanical ventilation (7).

Thoracic fluid content represents the whole (extravascular, intravascular, and intrapleural) fluid component in the thorax; thus, TFC was considered to provide an estimation of the extravascular lung water in absence of significant pleural or pericardial effusion (8,9).

Trans-thoracic echocardiography is a non-invasive tool that delivers bedside cardiac function evaluation. Echocardiography is now widely used to evaluate cardiac function during the ventilator weaning process. Impaired left ventricular systolic and diastolic function were reported to be good predictors of weaning failure (10).

Inferior vena cava (IVC) size and collapsibility can give us an idea about hypovolemic patients for estimation of right atrial pressure. Inferior vena cava diameter can be measured using the trans-thoracic echo-cardio graphic subcostal window in the sagittal plane. M-mode imaging allows high-frame rate measurements of size changes throughout the respiratory cycle (11).

Trans-mitral to mitral annular early diastolic velocity ratio (E/Ea ratio) is an echo Doppler non invasive estimation of left ventricular filling pressures and can be measured using trans-thoracic echo-cardiograph in the apical four-chamber view then pulse-wave Doppler imaging is done to record trans-mitral and mitral annular flow in early diastole (12).

DETAILED DESCRIPTION:
Rational Weaning of patients from mechanical ventilation is a critical problem in intensive care unit to prevent complications of prolonged intubation and ventilation of critically ill patients.

This pushes us to conduct this study to assess efficiency of measuring thoracic fluid content and Fluid Balance and some echo-cardio graphic parameters such as inferior vena cava maximum diameter (IVC max) and trans-mitral to mitral annular early diastolic velocity ratio (E/Ea ratio) as non invasive measures in predicting failed weaning from mechanical ventilation to reduce these hazards on the patients.

Research Question Is usage of non invasive measures as thoracic fluid content, Fluid balance, IVC max and E/Ea ratio beneficial in predicting failed weaning from mechanical ventilation in critically ill patients? Hypotheses

Null hypothesis (H0):

Thoracic fluid content measurement is not a good predictor For weaning from mechanical ventilation in critically ill patients.

Alternative hypothesis (H1):

Thoracic fluid content measurement is a good predictor for weaning from mechanical ventilation in critically ill patients.

Aim of the work Usage of Non invasive parameter for prediction of failed weaning from mechanical ventilation to prevent hazards of prolonged intubation and ventilation and to improve outcome in these critically ill patients.

Objectives To assess validity of Thoracic fluid content measurement, Fluid Balance, IVC max and E/Ea ratio as noninvasive parameters in predicting failed weaning from mechanical ventilation.

To compare efficiency of Thoracic fluid content measurement, Fluid Balance, IVC max and E/Ea ratio as noninvasive parameters in predicting failed weaning from mechanical ventilation.

To Examine the relationship of Thoracic fluid content measurement, Fluid Balance, IVC max and E/Ea ratio as noninvasive parameters and weaning outcomes.

Patients and Methods

Technical design:

Site of the study:

This study will be carried out in the Intensive care unit of Anesthesia, Intensive Care and Pain Management, Zagazig University Hospitals.

Duration of Study over three months. Type of study : prospective observational study.

Sample Size :

120 participant Patients included in this study

Inclusion criteria:

Patients or first degree relative's acceptance. All patients who are mechanically ventilated for more than 48 hours. Both sexes. Age: above 18 years old. Critically ill patients who suffer from multisystem diseases that can result in significant morbidity or mortality.

Exclusion criteria:

Patients with significant pleural or pericardial effusion. Presence of pneumothorax or severe subcutaneous emphysema. Patients with significant valvular heart lesions or atrial fibrillation. Patients with injuries or wounds which hinder application of device electrodes. Presence of burns at site of application of electrodes.

Operational design:

Parameters of the study:

Assessment for weaning readiness:

The decision of readiness to wean is performed by the attending ICU physician according to ICU protocol which includes these criteria (14) :

Improvement or resolution of the primary cause of intubation and ventilation. Presence of adequate cough power. Absence of excessive endobronchial secretions. Adequate oxygenation : PaO2 >60 mmHg or SpO2 >90% on FiO2 40% or less or PaO2/FiO2 ratio >150 .

Patient is not tachypneic where respiratory rate less than 30 breath per minute.

Stable cardiovascular state as regarding blood pressure and heart rate without active ischemia, high vasopressors or inotropic support .

No need for heavy sedation . Patient can initiate respiratory effort by himself. Absence of high fever or severe anemia. Prepare patient for weaning : proper positioning of the patient and suction of secretions and optimization of the circumstances.

Start weaning using spontaneous breathing trial (SBT): we set the ventilator to spontaneous pressure support mode with least parameters as poitive end expiratory pressure PEEP of 5 cmH2o and pressure support of 5-8 cmH2o with FiO2 40%. SBT will be continued for 30 minutes. Rapid shallow breathing index RSBI is calculated by dividing respiratory rate over tidal volume and then the patient is assessed for weaning criteria again to complete weaning from mechanical ventilation (15).

The decision of extubation is also performed by the attending ICU physician after fulfillment of extubation criteria which include adequate cough power, absence of airway edema, reasonable conscious level and performing cuff leak test.

Weaning failure is defined as re-intubation within 48 hours after extubation due the presence of one or more of the following criteria: tachypnea (respiratory rate more than 35 breaths per minute), oxygen saturation less than 90% or PaO2 less than 60 mmHg on a fraction of inspired oxygen of 40%, apparent increase in accessory respiratory muscle activity, and evident facial signs of respiratory distress (16).

Thoracic fluid content (TFC) is measured 5 minutes before SBT using electrical cardiometry device (ICONR monitor: Osypka Medical, Inc., La Jolla, California and Berlin). The ICON device is connected to four electrocardiogram electrodes which are placed over patients' skin after cleaning with alcohol at the neck below the left ear, just above the left clavicular midpoint, and two electrodes at left mid-axillary line one at the level of the xiphoid process, and the other electrode 5 cm below this point. The TFC is observed for 30 s and the average of the highest and lowest values is recorded with normal value ranges from 20 to 45 kΩ-1 (13).

Fluid balance 24 hours before SBT: (including fluids, medications and blood products) refers to inputs minus outputs (tallied at midnight) of the day prior to the SBT and days of mechanical ventilation will also be recorded. (17,18) Trans-thoracic echo-cardiographic data as IVCmax and E/Ea ratio are measured using the trans-thoracic echo-cardiographic subcostal window in the sagittal plane by angling and rotating the transducer to the left from the subcostal four-chamber (4C) view. M-mode imaging allows high-frame rate measurements of size changes throughout the respiratory cycle 5 minutes before performing SBT (12).

Hemodynamic data: systolic blood pressure and heart rate will be recorded 5 minutes before SBT.

All Patients are divided into successful weaning group and failed weaning group. Both groups are compared according to the study outcomes.

Collecting data:

From each patient the following data will be collected:

Patient characteristics (name, age, gender, body mass index (BMI)). Cause of intubation and mechanical ventilation. Date of ICU admission and cause of admission. Medical and past history. History of ICU admission before. Thoracic fluid content measurement. Fluid balance of the patient. Echo-cardiographic data as IVCmax and E\Ea ratio Hemodynamic data as systolic blood pressure and heart rate Duration of mechanical ventilation.

Administrative design:

Approval will be obtained from ethics committee of approval of the department of anesthesia and surgical intensive care.

Approval will be obtained from the Institutional review board (IRB) of faculty of medicine, zagazig university.

A Written Informed consent will be signed from all patients or first degree relatives will be obtained.

Results:

Collected data will be tabulated in tables and suitable graphs and analyzed according to standard statistical methods.

Discussion:

Discussion will be done on results compared to related relevant literature and scientific researches.

Conclusion & Recommendations:

will be derived from the findings of the study. References Boles J, Bion J., Connors A., Herridge M., Marsh B., Melot C., et al. (2007): Weaning from mechanical ventilation. Eur Respir J.; 29(1):1033-56.

Schmidt G.A., Girard T.D., Kress J.P., Morris P.E., Ouellette D.R., Alhazzani W., et al. (2017): Liberation from mechanical ventilation in critically ill adults: executive summary of an official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline. Chest.;151(1):160-5.

Frutos-Vivar F, Ferguson ND, Esteban A, Epstein SK, Arabi Y, Apezteguía C, et al. (2006): Risk factors for extubation failure in patients following a successful spontaneous breathing trial. Chest.;130(1):1664-71.

Frutos-Vivar F., Esteban A., Apezteguia C., González M., Arabi Y., Restrepo M.I., et al. (2011): Outcome of reintubated patients after scheduled extubation. J Crit Care.;26:502-9.

Dres M., Teboul J-L. and Monnet X. (2014): Weaning the cardiac patient from mechanical ventilation. Curr Opin Crit Care.;20(1):493-8.

Upadya A., Tilluckdharry L., Muralidharan V., Amoateng-Adjepong Y. and Manthous C.A. (2005): Fluid balance and weaning outcomes. Intensive Care Med.;31(1):1643-7.

Caille V., Amiel J-B., Charron C., Belliard G., Vieillard-Baron A. and Vignon P. (2010): Echocardiography: a help in the weaning process. Crit Care.;14(1): 120.

Narula J., Kiran U., Malhotra Kapoor P., Choudhury M., Rajashekar P. and Kumar C.U. (2017): Assessment of changes in hemodynamics and intrathoracic fluid using electrical cardiometry during autologous blood harvest. J Cardiothorac Vasc Anesth.;31 (1):84-9.

Hammad Y., Hasanin A., Elsakka A., Refaie A., Abdelfattah D., Rahman S.A., et al. (2019): Thoracic fluid content: a novel parameter for detection of pulmonary edema in parturients with preeclampsia. J Clin Monit Comput.;33(1):413- 8.

Almeida C.A., Nedel W.L., Morais V.D., et al. (2016): Diastolic dysfunction as a predictor of weaning failure: a systematic review and meta-analysis. J Crit Care.; 34: 135- 41.

Machare-Delgado E., Decaro M. and Marik PE. (2011): Inferior vena cava variation compared to pulse contour analysis as predictors of fluid responsiveness: a prospective cohort study. J Int Care Med.;26(1):116-24.

Rudski L.G., Lai W.W., Afilalo J., Hua L., Handschumacher M.D., Chandrasekaran K., et al. (2010): Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography. Endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr.;23(1):685-713.

Fathy Sh., Hasanin A., Raafat M., Mostafa M.A., Fetouh A.M., Elsayed M., et al. (2020): Thoracic fluid content: a novel parameter for predicting failed weaning from mechanical ventilation.Journal of intensive car.;8(1): 20-1.

Karthika M., Al Enezi F., Pillai L., et al. (2016): Rapid shallow breathing index. Ann Thorac Med., 11(3):167- 76.

Peñuelas Ó., Thille A.W. and Esteban A. (2015): Discontinuation of ventilatory support. Curr Opin Crit Care.;21(1):74-81.

Epstein SK, Ciubotaru RL and Wong JB. (1997): Effect of failed extubation on the outcome of mechanical ventilation. Chest.;112(1):86-8.

Carolina A., Antonio P., Teixeira C., Castro PS., Savi A., Oliveira RP., Gazzana MB., et al. (2015): 48-Hour Fluid Balance Does Not Predict a Successful Spontaneous Breathing Trial. RESPIRATORY CARE; 60 (8): 1091- 2.

Upadya A., Tilluckdharry L.,Muralidharan V.,Yaw Amoateng-Adjepong Y. and Manthous C. (2005): Fluid balance and weaning outcomes. Intensive Care Med.; 31(1):1643- 7.

ELIGIBILITY:
Inclusion Criteria:

* 2. Patients or first degree relative's acceptance. All patients who are mechanically ventilated for more than 48 hours. 3. Gender: both sexes. 4. 5. Age: above 18 years old. Critically ill patients who suffer from multisystem diseases that can result in significant morbidity or mortality.

Exclusion Criteria:

- 1. Patients with significant pleural or pericardial effusion. 2. Presence of pneumothorax or severe subcutaneous emphysema. 3. Patients with significant valvular heart lesions or atrial fibrillation. 4. Patients with injuries or wounds which hinder application of device electrodes.

5. Presence of burns at site of application of electrodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient who are mechanically ventilated in ICU from both sex suffering from multi system process that may result in significant morbidity and mortality
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
To assess role of thorathic fluid content measurement by using cardiometry in weaning from mechanical ventilation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Sharqia Province, Egypt